CLINICAL TRIAL: NCT05649683
Title: Immunological Functionnal Test Validation to Predict Melanoma Metastatic Patient Response to Checkpoint Inhibitors - Melanoma Quantiferon
Brief Title: Immunological Functionnal Test Validation to Predict Melanoma Metastatic Patient Response to Checkpoint Inhibitors
Acronym: mela-quantif
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 22-PP-14
Record Dates: First submitted 2022-11-24; First posted 2022-12-14 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Melanoma (Skin)
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Analysis of blood cytokine (Other): Patients will receive anti-PD1 therapy (Nivolumab/Nivo) with anti-CTLA4 therapy (Ipilimumab/Ipi) as part of routine care, as per the MA scheme followed in case of efficacy and good tolerance of Nivolumab maintenance treatment alone. The functional test for cytokines (1ml total blood on lihtium heparinate) will be performed at the initiation of ICI (J0), at week 6 (S6, after the 2nd cure), at week 11 (S11= 1st radiological evaluation, after the 4 cures of Nivo+Ipi), and, if applicable, the progression of the disease and/or the occurrence of an ESi grade 3-4. Stimulated lymphocytes from non-therapy responders will be tested in vitro by various immunomodulatory drugs.
  During each sampling we will also collect 5 ml of serum on dry tube for serological constitution, 3ml on EDTA tube for performing an immunophenotyping (T, B, NK) and 3ml on EDTA tube for freezing total PBMC and setting up a biobank.
  Interventions: Biological: Evaluation of cytokine production

INTERVENTIONS:
Biological: Evaluation of cytokine production — The patient will have samples at initiation of treatment (J0), after treatments 1 and 2 (S6), after the first radiological assessment at S11 and/or the progression of the disease and/or occurrence of a grade 3-4 adverse event

SUMMARY:
Checkpoint inhibitor such as anti-CTLA-4 and anti-PD-1 are known to block inhibitory signals and increase the immune antimutoral response. Nivolumab and Ipilimumab association is considered as a more efficient immunotherapy to treat advanced melanoma. This combined immunotherapy is also responsible of severe immunes toxicyties. Identification of predictives biomarqueurs remains a challenge to predict the balance between tolerability and efficency. Previous data showed that advanced melanoma patient had lower level of Th1 cytokines that predict a less efficient immune system than healthy donors. The second point was that high level of Th1 and Th17 cytokines were correlate to a better tumor response. The last point was that patients with severe immune toxicity showed an increase of IL-6 and IL17a production. The investigators would like to identify the predictive values of Th1, Th2 and Th17 at the begining and during the combined immunotherapy and correlate these cytokines levels secretions to a potential efficient tumor response or to the emergence of induced immunes toxicities. This study is an original approach using functionnal test to predict the balance between efficienty and tolerability.

ELIGIBILITY:
Inclusion

* persone of major age,
* advanced melanoma confirmed,
* RECIST 1.1 disease,
* first line treatment

Exclusion Criteria:

* occular and mucosal melanoma,
* previous checkpoint inhibitor treatment,
* active brain metastasis,
* concomitant immunosuppressive treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-31 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of predictifve Th1, Th2 and Th17 cytokine production correlate to the RECIST 1.1 tumoral response | Change from Baseline tumoral response at week 6 and at week 11
  Analysis of blood cytokine secretion upon non specific in vitro stimulation RECIST 1.1 tumor response

SECONDARY OUTCOMES:
Evaluation of predictifve Th1, Th2 and Th17 cytokine production correlate to the progression free | Change from Baseline disease progression at week 6 and at week 11
  Analysis of blood cytokine secretion upon non specific in vitro stimulation disease progression
Evaluation of predictifve Th1, Th2 and Th17 cytokine production correlate to severe immunological toxicity occurrence | Change from Baseline immunological toxicity occurrence at week 6 and at week 11
  Analysis of blood cytokine secretion upon non specific in vitro stimulation severe immunological toxicity occurrence

CONTACTS AND LOCATIONS:
Overall Officials: Montaudie Henri, PhD, Principal Investigator — CHU de Nice, Service de Dermatologie
Locations (3):
- France (3):
  - CHU de Nice - Hôpital de l'Archet, Nice, Alpes-maritimes
  - CHU de Montpellier, Montpellier, Occitanie
  - CHRU de Lille, Lille

IPD SHARING:
Plan to Share IPD: No